CLINICAL TRIAL: NCT04163471
Title: VasoStat vs. TR Band for Hemostasis Following Transradial Catheterization Without Prior Radial Access
Brief Title: VasoStat vs. TR Band for Radial Hemostasis
Status: Completed | Type: Observational
Sponsor: Forge Medical (Industry)
Collaborators: Billings Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 20181194
Record Dates: First submitted 2018-08-22; First posted 2019-11-14 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: Coronary Artery Disease; Peripheral Arterial Disease
Keywords: VasoStat; TR Band; Transradial access; Coronary angiography; Peripheral arterial disease; Coronary artery disease; Peripheral angiography; Stents
MeSH Terms: conditions — Coronary Artery Disease; Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- VasoStat: Randomized to use of VasoStat radial mechanical compression for hemostasis device following sheath removal after transradial access for arterial catheterization procedures.
  Interventions: Device: Radial artery mechanical compression for hemostasis
- TR Band: Randomized to use of TR Band radial mechanical compression for hemostasis device following sheath removal after transradial access for arterial catheterization procedures.
  Interventions: Device: Radial artery mechanical compression for hemostasis

INTERVENTIONS:
Device: Radial artery mechanical compression for hemostasis — Transradial hemostasis following arterial catheterization procedures

SUMMARY:
VasoStat vs. TR Band compression for Radial Artery Hemostasis Following Transradial Catheterization Without Prior Radial Artery Access

DETAILED DESCRIPTION:
Patients will be enrolled if they are scheduled to undergo a coronary or peripheral catheterization procedure involving the placement of a sheath (plastic tube) in the radial artery near the participants wrist. The purpose of this research is to compare two devices which make bleeding stop after the participants procedure is finished and the plastic tube is removed from the radial artery in the wrist. The two devices are called the VasoStat and the TR Band. Both of these devices are called hemostasis devices, which means they stop bleeding (hemostasis). Both devices are approved by the Food and Drug Administration (FDA) and are used throughout hospitals in the United States. The investigators will compare blood flow to the hand, and survey patients as to how comfortable these devices are, while they are being used to stop bleeding after the catheterization procedure.

Patients will be randomized to one device or the other as part of the study.

The investigators will noninvasively measure the blood flow to the hand by placing a soft plastic probe on the tip of the thumb called a plethysmography probe. This measurement only takes a few seconds and is painless. The investigators will measure before, after application and after removal & before patients are discharged. Thirty days later, patients will return for another measurement and to examine the radial artery with an ultrasound probe.

40 patients will be enrolled. Statistical analysis: Based on prior studies, The investigators will assume that the VasoStat produces a 30% reduction in hand perfusion during normal clinical use. The investigators assume the TR Band produces a 70% reduction in hand perfusion during normal clinical use. Using a two-sample test of proportions, with a Type I error of 5%, a power of 80%, and an anticipated drop-out rate of 10%, The investigators will need to enroll 40 patients (20 patients in each arm of the study) (StatMate 2.0, GraphPad Software, San Diego, CA)

ELIGIBILITY:
Inclusion Criteria:

• no prior radial access

Exclusion Criteria:

* Patients receiving concurrent investigational medications
* Cellulitis overlying radial artery
* Oral anticoagulation
* Patients receiving glycoprotein IIb/IIIa inhibitors
* Dementia
* Prisoners
* Institutionalized individuals
* Allergy to medical adhesive
* Radial sheath > 6 French (ID)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients referred for diagnostic or interventional arterial catheterization procedures who have coronary artery disease or peripheral artery disease
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2019-03-06 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Comparison of impact of two radial artery compression devices on hand perfusion measurements | Perfusion index measurements day 1: before radial artery puncture, during wrist compression, after removal of compression device. Final perfusion index at 30-day followup appointment.
  Changes in Hand perfusion will be quantified using a noninvasive pulse oximetry technique and a previously validated metric known as the Perfusion Index, which is the ratio of the pulsatile blood flow to the nonpulsatile or static blood in peripheral tissue. The Perfusion Index represents a noninvasive measure of hand perfusion that can be continuously and noninvasively obtained from a specialized pulse oximeter.

SECONDARY OUTCOMES:
Comparison of impact of two radial artery compression devices on hand perfusion prior to and during ulnar artery compression | Perfusion index measurements on day 1 with ulnar compression: will include before radial artery puncture, and during wrist compression after radial sheath removal.
  Changes in Hand perfusion will be quantified using a noninvasive pulse oximetry technique and a previously validated metric known as the Perfusion Index, which is the ratio of the pulsatile blood flow to the nonpulsatile or static blood in peripheral tissue. The Perfusion Index represents a noninvasive measure of hand perfusion that can be continuously and noninvasively obtained from a specialized pulse oximeter.
Patient satisfaction during use of wrist compression device | During application of radial artery mechanical compression
  Survey of patient perception of wrist discomfort, hand numbness, pain, swelling and willingness to use again in the future
Hand perfusion and radial artery patency after one month | 30 day follow-up after use of mechanical wrist compression following transradial access for arterial catheterization procedures
  Changes in Hand perfusion will be quantified using a noninvasive pulse oximetry technique and a previously validated metric known as the Perfusion Index, which is the ratio of the pulsatile blood flow to the nonpulsatile or static blood in peripheral tissue. The Perfusion Index represents a noninvasive measure of hand perfusion that can be continuously and noninvasively obtained from a specialized pulse oximeter. Duplex ultrasound will be used to assess radial artery patency.

OTHER OUTCOMES:
Adverse outcomes | During index hospital visit and at 30 day follow-up
  Hematoma, swelling, pain, paresthesia, arterial venous fistula, pseudoaneurysm, partial or total radial artery occlusion

CONTACTS AND LOCATIONS:
Locations (1):
- Billings Clinic Heart and Vascular at Community Medical Center, Missoula, Montana, United States

IPD SHARING:
Plan to Share IPD: Undecided